CLINICAL TRIAL: NCT04975451
Title: Neoadjuvant Treatment Anlotinib Combined With Docetaxel and Carboplatin in Triple-negative Early-stage Breast Cancer : a Multicenter, Open, Single-arm Phase II Trial
Brief Title: ADCb (Anlotinib/Docetaxel/Carboplatin) as Neoadjuvant Therapy for Triple-Negative Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Anqin Zhang (Other)
Responsible Party: Sponsor-Investigator, Anqin Zhang, Chief Physician, Guangdong Women and Children Hospital
Organization: Guangdong Women and Children Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GDWCH002(TNBC)
Record Dates: First submitted 2021-07-14; First posted 2021-07-23 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ADCb (Experimental): Anlotinib (anlotinib 12mg qd p.o. d1-14/21day/cycle)and Docetaxel (75 mg/m2 administered intravenously every 3 weeks) and carboplatin (area under the concentration-time curve [AUC] 6, intravenously every 3 weeks) for six cycles
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — Anlotinib plus DCb

SUMMARY:
DCb (docetaxel/carboplatin) regimens as Neoadjuvant Treatment for Triple-Negative Breast Cancer have been recommended by NCCN guideline.Combination of anti-angiogenesis inhibitors is expected to further improvePathologic Complete Response(PCR).This study is to evaluate the efficacy and safety of ADCb (Anlotinib/docetaxel/carboplatin) as Neoadjuvant Treatment in Triple-Negative breast cancer. The endpoint of PCR is used as a surrogate marker for survival. Safety and tolerability assessed by number of grade 4 toxicities and hospitalizations.

DETAILED DESCRIPTION:
Triple negative breast cancer (TNBC) accounts for 15-20% of all invasive breast cancer,it is a subtype lacking estrogen receptor (ER), progesterone receptor (PR) and human epidermal growth factor receptor type 2 (HER2) amplification. The mainstay of treatment for TNBC is cytotoxic chemotherapy. However, despite its sensitivity to chemotherapy, TNBC is still associated with a poor prognosis and a higher risk of visceral transfer.

The benefits of neoadjuvant therapy include reducing the size of the tumor to suit breast conserving surgery, avoiding axillary lymph node dissection, making inoperable tumors operable, and obtaining an in vivo evaluation of the tumor's chemosensitivity.TNBC is usually recommended for neoadjuvant therapy. Taxane- and anthracycline-based neoadjuvant regimens have become a standard treatment for TNBC, and patients have been proved to have better event-free survival (EFS) and overall survival (OS) who achieve a pathologic complete response (pCR) after neoadjuvant chemotherapy.Previous studies have shown that adding carboplatin to neoadjuvant chemotherapy regimens significantly improved pCR rate in TNBC patients.The use of immunotherapy, parp inhibitors, and anti-angiogenesis inhibitors can improve PCR for triple-negative breast cancer neoadjuvant therapy.

This study was designed to see the efficacy and safety of Anlotinib plus docetaxel and carboplatin Neoadjuvant Treatment for Triple-Negative Breast Cancer.

ELIGIBILITY:
Inclusion Criteria：

1. Female, aged 18 Years to 75 Years
2. Signed written informed consent approved by the study site Ethics Committee
3. Histologically confirmed Triple-Negative invasive breast carcinoma：Pathologically confirmed as triple negative, defined as ER and PR expression both < 1 % of tumor cell nuclei per ASCO/CAP guidelinesa and HER2 negative per ASCO/CAP guidelinesa (IHC 0 or 1+ or FISH-, or IHC 2+ and FISH-)
4. Stage at presentation: II - III (T1cN1-2 or T2-4N0-2)
5. Patients must have measurable disease as defined by palpable lesion with caliper and/or a positive mammogram or ultrasound. Bilateral mammogram is required for study entry. Baseline measurements of the indicator lesions must be recorded on the Patient Registration Form. To be valid for baseline, the measurements must have been made within the 14 days if palpable. If not palpable, a mammogram or MRI must be done within 14 days. If palpable, a mammogram or MRI must be done within 2 months prior to study entry. If clinically indicated, x-rays and scans must be done within 28 days of study entry.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1 within 14 days of study entry
7. Adequate organ function within 2 weeks of study entry:
8. ANC ≥ 1500 cells/μL Platelet count ≥ 100,000 cells/μL Hemoglobin ≥ 9 g/dL; patients may receive red blood cell transfusions to obtain this level Serum creatinine ≤ 1.5 × upper limit of normal (ULN) INR and (activated) partial thromboplastin time (aPTT/PTT) ≤ 1.5 ×ULN AST and ALT ≤ULN Serum total bilirubin ≤ ULN, except for patients with Gilbert's syndrome for whom direct bilirubin should be within the normal range Serum alkaline phosphatase ≤ULN
9. Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment
10. Women of childbearing potential must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation

Exclusion Criteria:

1. Stage IV (metastatic) breast cancer
2. Patients with a history of invasive breast cancer.
3. Patients with a history of ductal carcinoma in situ (DCIS), except for patients treated exclusively with mastectomy > 5 years prior to diagnosis of current breast cancer
4. Patients with bilateral breast cancer
5. Prior chemotherapy, hormonal therapy, biologic therapy, investigational agent, targeted therapy or radiation therapy for current breast cancer.
6. Patients who have undergone incisional and/or excisional biopsy of primary tumor and/or axillary lymph nodes
7. History of previous or current malignancy at other sites with the exception of adequately treated carcinoma in-situ of the cervix or basal or squamous cell carcinoma of the skin. Patients with a history of other malignancies, who remain disease free for greater than five years are eligible.
8. Current severe, uncontrolled systemic disease that may interfere with planned treatment (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease; wound-healing disorders)
9. Major surgical procedure unrelated to breast cancer or significant traumatic injury within 28 days prior to randomization or anticipation of the need for major surgery during the course of study treatment
10. Current pregnancy and/or breastfeeding

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response(PCR) | Up to approximately 20-25 weeks
  Local evaluation of pCR defined as the absence of any residual invasive cancer of the resected breast specimen and all sampled ipsilateral lymph nodes (i.e., ypT0/is, ypN0 in the current AJCC staging system

SECONDARY OUTCOMES:
event-free survival(EFS) | Up to approximately 24 months
  defined as time from randomization to disease progression, disease recurrence (local, regional, distant, or contralateral [invasive or non-invasive]), or death from any cause
Safety and Tolerability | Up to approximately 20-25 weeks
  Incidence, type, and severity of all adverse events (including serious adverse events) based on NCI CTCAE, v4.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Women and Children Hospital, Guangzhou, Guangdong, China